CLINICAL TRIAL: NCT01542489
Title: An Observational 3 Months Study to Evaluate the Effect of Insulin Levemir® on Glycaemic Control, Weight and Incidence of Hypoglycaemic Events in Insulin Treated Subjects With Type 1 or Type 2 Diabetes
Brief Title: Observational Study of the Predictability of Levemir® in Terms of Metabolic Control, Change of Body Weight and Hypos
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN304-1927
Record Dates: First submitted 2012-02-24; First posted 2012-03-02 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir; Insulin Aspart

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- IDet + IAsp users
  Interventions: Drug: insulin detemir; Drug: insulin aspart
- IDet + HI users
  Interventions: Drug: insulin detemir; Drug: human soluble insulin

INTERVENTIONS:
Drug: insulin detemir — Prescribed by the physician solely as a result of a normal clinical evaluation. The physician determines the starting dose and frequency, as well as later changes to either dose or frequency, if any
Drug: insulin aspart — Prescribed by the physician solely as a result of a normal clinical evaluation. The physician determines the starting dose and frequency, as well as later changes to either dose or frequency, if any
  Groups: IDet + IAsp users
Drug: human soluble insulin — Prescribed by the physician solely as a result of a normal clinical evaluation. The physician determines the starting dose and frequency, as well as later changes to either dose or frequency, if any
  Groups: IDet + HI users

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to evaluate the effect of Levemir® (insulin detemir) on glycaemic control, weight and incidence of hypoglycaemic events in insulin treated subjects with type 1 or type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Any subject with type 1 or type 2 diabetes treated with insulin in whom at the discretion of the participating physicians it was decide to switch insulin treatment to the long-acting insulin analogue insulin detemir (Levemir®) in combination with either insulin aspart (NovoRapid®) or human insulin (Actrapid®)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any subject with type 1 or type 2 diabetes treated with insulin in whom at the discretion of the participating physicians it was decide to switch insulin treatment to the long-acting insulin analogue Levemir® in combination with either insulin aspart (NovoRapid®) or human insulin (Actrapid®)
Sampling Method: Non-Probability Sample
Enrollment: 480 (Actual)
Dates: Start 2006-10; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c (glycosylated haemoglobin)

SECONDARY OUTCOMES:
Change in 7-point blood glucose variability
Change in body weight
Insulin dose
Number of injections
Number of hypoglycaemic episodes
Number of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Bratislava, Slovakia

REFERENCES:
- [Result] Emil Martinka; Improved Glycemic Control and Weight Loss in Slovakian Patients Switching from NPH to Insulin Detemir; 2049-PO; 69th Scientific Sessions (2009); American Diabetes Association
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com